CLINICAL TRIAL: NCT05116995
Title: Differential EFfects of Dual antIplatelet and Dual aNtithrombotic thErapy on Hemostasis in Chronic Coronary Syndrome Patients: Define CCS Study, a Prospective Randomized Crossover Clinical Trial.
Brief Title: Differential EFfects of Dual antIplatelet and Dual aNtithrombotic thErapy on Hemostasis in Chronic Coronary Syndrome Patients
Acronym: DEFINE CCS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Wael Sumaya, Interventional Cardiologist, Nova Scotia Health Authority
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SUM001
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Thrombosis; Myocardial Infarction
MeSH Terms: conditions — Thrombosis; Myocardial Infarction | interventions — Rivaroxaban; Ticagrelor

STUDY DESIGN:
Intervention Model Description: Treatment #1 for one week then on Day 21 they enter Treatment #2 for 1 week.
Who Masked: Care Provider
Masking Description: Study personnel performing bleeding time and laboratory staff will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban first (Active Comparator): Patients will be treated with rivaroxaban 2.5 mg twice a day for one week then on Day 21, will be treated with ticagrelor 60 mg twice a day for one week.
  Interventions: Drug: Rivaroxaban; Drug: Ticagrelor
- Ticagrelor first (Active Comparator): Patients will be treated with ticagrelor 60 mg twice a day for one week then on Day 21, will be treated with rivaroxaban 2.5 mg twice a day for one week.
  Interventions: Drug: Rivaroxaban; Drug: Ticagrelor

INTERVENTIONS:
Drug: Rivaroxaban — rivaroxaban 2.5 mg twice a day for 7 days
  Other Names: xarelto
Drug: Ticagrelor — Ticagrelor 60 mg twice a day for 7 days
  Other Names: brilinta

SUMMARY:
The investigators will be comparing the effects of two different drug treatment strategies, in patients with history of a heart attack, on different markers of bleeding and clotting risk. Both treatment strategies are already approved for the indication of improving outcomes in high-risk patients with history of heart attack.

DETAILED DESCRIPTION:
The investigators will enroll patients with coronary disease >1 year after an acute coronary syndrome. Subjects will be randomized to one of two treatment plans. One plan the participant will take ticagrelor for one week, then take two weeks off with no drug (washout period), then one week of rivaroxaban. The other plan will be reverse order where the participant will take rivaroxaban for one week, then two weeks off(washout period), then one week of ticagrelor. Study drugs will be provided to participants at the start of each treatment period. Bleeding time will be determined and blood samples will be taken at four timepoints (baseline, post first drug, pre second drug, and post second drug) to measure complete blood count, CRP, and fibrin clot assessment. These are surrogate markers for safety (bleeding) and efficacy (increased thrombotic risk)

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic coronary syndrome (at least 1 year after having a myocardial infarction) on aspirin monotherapy will be eligible for this study. They have to have at least one of these additional risk factors:

  1. Diffuse coronary artery disease.
  2. Peripheral vascular disease
  3. Diabetes
  4. Chronic kidney disease (eGFR<60 ml/unit/1.73 m2)

Exclusion Criteria:

* Allergy to either rivaroxaban or ticagrelor
* Requirement for anticoagulation or P2Y12 inhibitor therapy
* Anemia (hemoglobin < 10 g/dL)
* Severe renal impairment (eGFR < 30 ml/unit/1.73 m2)
* Bleeding disorders
* Significant liver impairment resulting in deranged clotting parameters
* Any history of intracranial hemorrhage
* Stroke within 6 months
* History of gastrointestinal bleed within 6 months
* Major surgery within 1 month
* Patients with inflammatory conditions
* Concomitant treatment with immunosuppressive therapy, inhibitors or inducers of P glycoprotein or CYP3A4 enzymes (eg. azole antifungals, ritonavir, erythromycin, clarithromycin, rifampicin)
* Concomitant treatment with antidepressants (selective serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors)
* Pregnancy
* Inability to give written consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding time | 7 days
  The primary objective is to determine the differential effect of rivaroxaban and ticagrelor on bleeding time as a surrogate marker for bleeding tendency.

SECONDARY OUTCOMES:
Differential effects on inflammatory markers (white cell count and CRP) | 7 days
  These will be measured from blood draws
Differential effects on fibrin clot lysis time | 7 days
  This will be measured from blood draws

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No